CLINICAL TRIAL: NCT02332564
Title: Coronary Steal Via Natural Internal Mammary Artery-To-Coronary Artery Bypasses
Acronym: CIMA
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SNCTP000001138; 2631 (Other: Bern University Hospital)
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Ischemia
Keywords: Circulation, Collateral; Coronary Artery Disease; Internal Mammary-Coronary Artery Anastomosis; Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Coronary Artery Disease: Patient with significant coronary artery disease
  Interventions: Other: Coronary Artery Balloon Occlusion for Determination of Collateral Flow Index
- No Coronary Artery Disease: Patient without significant coronary artery disease
  Interventions: Other: Coronary Artery Balloon Occlusion for Determination of Collateral Flow Index

INTERVENTIONS:
Other: Coronary Artery Balloon Occlusion for Determination of Collateral Flow Index — Coronary Artery Balloon Occlusion for Determination of Collateral Flow Index

SUMMARY:
CORONARY ARTERY DISEASE AND THE BENEFIT OF BYPASSES

Despite considerable advances in medicine, cardiovascular diseases remain the number one cause of death globally. In industrialized countries, coronary artery disease (CAD) is the leading cause of death, consequence of myocardial infarction (MI). Artificial - or natural - bypasses exert a protective effect by providing an alternative source of blood flow to a myocardial territory potentially affected by an acute coronary occlusion. Coronary collaterals represent pre-existing inter-arterial anastomoses and as such are the natural counter-part of surgically created bypasses. In patients with chronic CAD, sufficient coronary collaterals have been shown to confer a significant benefits in terms of overall mortality and cardiovascular events.

EXTRACARDIAC-TO-CORONARY COLLATERAL SUPPLY

Commonly, coronary collaterals are implicitly understood to exist between coronary artery branches. However, the structural existence of coronary collaterals with an extracardiac connection has been confirmed by anatomical investigations. Pathophysiologically and with regard to a potential for arteriogenic stimulation, the connections from the internal mammary arteries, are of special interest.

In a recently published work the investigators have investigated the effect of temporary balloon occlusion of the distal IMA on coronary collateral function. There were equivocal findings for the left circumflex coronary artery: CFI was increased by ipsilateral IMA occlusion, but the level of myocardial ischemia was unchanged.

MYOCARDIAL STEAL VIA INTERNAL MAMMARY ARTERIES

In the investigators' previous study, the coronary occlusion with simultaneous distal IMA occlusion was always performed first as a conservative measure against false-positive detection of internal-mammary-to-coronary artery connections. Repetitive coronary occlusions per se result in higher collateral flow by collateral recruitment and reduced ischemia by ischemic preconditioning and augmented collateral function. Conversely, the sensitivity of the employed method was reduced and might have contributed to the equivocal findings in case of the left circumflex artery. Moreover, the hypothesize d mechanism of localized pressure augmentation was not investigated.

This study aims to further characterize the prevalence and function of natural ipsilateral IMA-to-coronary connections, as well as to investigate the hemodynamic mechanisms of coronary collateral function augmentation by distal IMA occlusion. In the investigators' last study, the increased coronary collateral function in response to manipulation of a potential coronary collateral donor (in this case, the IMA) was taken as indirect evidence for the existence of IMA-to-coronary-artery connections. Thus, the employed distal IMA occlusion served as a positive stimulus. Conceptually, additional evaluation with a negative stimulus could heighten the discriminatory power of the investigation. This could be in the form of a hyperemic stimulus affecting the collateral donor, ie in analogy to myocardial or coronary steal (ie, a reduction in coronary collateral supply to a collateral recipient).

DETAILED DESCRIPTION:
CORONARY ARTERY DISEASE AND THE BENEFIT OF BYPASSES

Despite considerable advances in medicine, cardiovascular diseases remain the number one cause of death globally. In industrialized countries, coronary artery disease (CAD) is the leading cause of death, consequence of myocardial infarction (MI).

In patients with acute coronary syndrome, percutaneous coronary intervention (PCI) has been shown to improve outcomes.2 However, in stable CAD, PCI has not been demonstrated to reduce the incidence of myocardial infarction or death. Coronary artery bypass grafting (CABG) was superior to PCI in patients with diabetes and multivessel coronary artery disease. CABG significantly reduced rates of death and myocardial infarction compared to PCI, but with a higher rate of stroke. Furthermore, in patients with advanced coronary artery disease, rates of myocardial infarction were more than 60% lower with CABG compared to PCI.

Conceptually, the benefit of CABG over PCI is not surprising as PCI targets significant coronary lesions thought to be responsible for causing ischemia. However, the deleterious effects of atherosclerosis are not typically preceded by significant luminal vascular narrowing. The vulnerable plaque eventually becoming the culprit plaque (causing myocardial infarction or sudden cardiac death) is typically relatively nonstenotic. Furthermore, due to being multifocal and widespread, plaque vulnerability is not a target for, nor amenable to PCI.

Conversely, artificial - or natural - bypasses exert a protective effect by providing an alternative source of blood flow to a myocardial territory potentially affected by an acute coronary occlusion. Coronary collaterals represent pre-existing inter-arterial anastomoses and as such are the natural counter-part of surgically created bypasses. In patients with chronic CAD, sufficient coronary collaterals have been shown to confer a significant benefits in terms of overall mortality and cardiovascular events.

EXTRACARDIAC-TO-CORONARY COLLATERAL SUPPLY

Commonly, coronary collaterals are implicitly understood to exist between coronary artery branches. However, the structural existence of coronary collaterals with an extracardiac connection has been confirmed by anatomical investigations. Pathophysiologically and with regard to a potential for arteriogenic stimulation, the connections from the internal mammary arteries, are of special interest. Indeed, before the advent of coronary bypass surgery, several clinical studies examined the usefulness of a minimally invasive surgery to augment collateral flow to the heart via these internal-mammary-to-coronary-artery connections in patients with angina pectoris. The performed distal bilateral ligation of the internal mammary arteries was thought to improve flow over naturally pre-existing anastomoses between the internal mammary arteries and the coronary circulation.

In a recently published work the investigators have investigated the effect of temporary balloon occlusion of the distal IMA on coronary collateral function. 180 pairs of measurements were performed in 120 patients electively referred for coronary angiography. Levels of collateral function and myocardial ischemia were determined during two coronary balloon occlusions, the first with, the second without distal IMA balloon occlusion. Coronary collateral function, determined by collateral flow index (CFI) was consistently increased by ipsilateral, but not contralateral IMA balloon occlusion in the left anterior descending (LAD) coronary artery and the right coronary artery (RCA). Furthermore, these findings were corroborated by the observed reduction in ischemia as assessed by the sensitive tool of intracoronary ECG. However, there were equivocal findings for the left circumflex coronary artery: CFI was increased by ipsilateral IMA occlusion, but the level of myocardial ischemia was unchanged.

MYOCARDIAL STEAL VIA INTERNAL MAMMARY ARTERIES

In the investigators' previous study, the coronary occlusion with simultaneous distal IMA occlusion was always performed first as a conservative measure against false-positive detection of internal-mammary-to-coronary artery connections. Repetitive coronary occlusions per se result in higher collateral flow by collateral recruitment and reduced ischemia by ischemic preconditioning and augmented collateral function. Conversely, the sensitivity of the employed method was reduced and might have contributed to the equivocal findings in case of the left circumflex artery. Moreover, the hypothesize d mechanism of localized pressure augmentation was not investigated.

This study aims to further characterize the prevalence and function of natural ipsilateral IMA-to-coronary connections, as well as to investigate the hemodynamic mechanisms of coronary collateral function augmentation by distal IMA occlusion. In the investigators' last study, the increased coronary collateral function in response to manipulation of a potential coronary collateral donor (in this case, the IMA) was taken as indirect evidence for the existence of IMA-to-coronary-artery connections. Thus, the employed distal IMA occlusion served as a positive stimulus. Conceptually, additional evaluation with a negative stimulus could heighten the discriminatory power of the investigation. This could be in the form of a hyperemic stimulus affecting the collateral donor, ie in analogy to myocardial or coronary steal (ie, a reduction in coronary collateral supply to a collateral recipient).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Referred for elective coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria:

* Acute coronary syndrome; unstable cardiopulmonary conditions
* Severe cardiac valve disease
* Congestive heart failure NYHA III-IV
* Prior coronary artery bypass surgery / prior cardiac surgery
* Coronary artery disease unsuitable for intracoronary pressure measurements
* Prior Q-wave myocardial infarction in the vascular territory undergoing collateral function determination
* Severe renal or hepatic failure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients electively referred for coronary angiography
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2020-11 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Coronary collateral function (CFI) | Baseline
  Coronary collateral function (CFI)

SECONDARY OUTCOMES:
Myocardial ischemia during temporary coronary balloon occlusion | Baseline
Proximal IMA pressure immediately before and during (ipsilateral) reactive arm hyperemia. | Baseline
Distal IMA CFI | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof., Principal Investigator — Department of Cardiology, Bern University Hospital
Locations (1):
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Stoller M, de Marchi SF, Seiler C. Function of natural internal mammary-to-coronary artery bypasses and its effect on myocardial ischemia. Circulation. 2014 Jun 24;129(25):2645-52. doi: 10.1161/CIRCULATIONAHA.114.008898. Epub 2014 Apr 17. PMID 24744276
- [Background] BLAIR CR, ROTH RF, ZINTEL HA. Measurement of coronary artery blood-flow following experimental ligation of the internal mammary artery. Ann Surg. 1960 Aug;152(2):325-9. doi: 10.1097/00000658-196008000-00018. No abstract available. PMID 13801236
- [Background] Bigler MR, Buffle E, Stoller M, Grossenbacher R, Tschannen C, Seiler C. Extracardiac coronary steal induced by upper limb hyperemia: a feature of internal mammary artery arteriogenesis. J Appl Physiol (1985). 2021 Sep 1;131(3):905-913. doi: 10.1152/japplphysiol.00082.2021. Epub 2021 Jul 8. PMID 34236245